CLINICAL TRIAL: NCT00233610
Title: A Comparative Trial of the Efficacy of Two Different Nolvadex (NDX) Dosing and Scheduling Regimens in Preventing Gynecomastia Induced by Casodex (CDX) 150 Monotherapy in Prostate Cancer Patients. An Open, Multicenter, Phase III Trial.
Brief Title: Two Different Regimens of Nolvadex in Preventing Gynecomastia Induced by Casodex 150 mg in Patients With Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 7054IT/0003
Record Dates: First submitted 2005-10-04; First posted 2005-10-06 (Estimated); Last update posted 2011-01-27 (Estimated); Status verified 2011-01

CONDITIONS: Prostate Cancer
Keywords: Casodex monotherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; Tamoxifen

INTERVENTIONS:
Drug: Bicalutamide
Drug: Tamoxifen

SUMMARY:
The aim of the study is to investigate the efficacy of different dosing and scheduling of Nolvadex in preventing gynecomastia/mastalgia induced by Casodex 150 mg monotherapy in patients with prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate cancer
* Locally advanced prostate cancer patients suitable for Casodex 150 mg monotherapy

Exclusion Criteria:

* Age > 75 yrs
* No metastatic disease (M1).
* No presence of gynaecomastia and/or mastalgia at screening
* No therapy with medications able to provoke gynaecomastia and/or mastalgia within 6 months of trial entry.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 2003-12; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Incidence of Gynecomastia and Breast pain at 2, 6 months and every 6 months thereafter and/or at withdrawal visit.

SECONDARY OUTCOMES:
Sexual functioning, Quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Astra Zeneca, Study Director — AstraZeneca
Locations (11):
- Italy (11):
  - Research Site, Bari, BA
  - Research Site, Bologna, BO
  - Research Site, Catania, CT
  - Research Site, Bagno a Ripoli, FI
  - Research Site, Florence, FI
  - Research Site, Genova, GE
  - Research Site, Pisa, PI
  - Research Site, Parma, PR
  - Research Site, Roma, Roma
  - Research Site, Udine, UD
  - Research Site, Como